CLINICAL TRIAL: NCT03250039
Title: A Phase 1, Open-label, Non-randomized, 2-period, Fixed Sequence Study To Investigate The Absorption, Metabolism And Excretion Of [14c-pf-04965842] And To Assess The Absolute Bioavailability And Fraction Absorbed Of Pf-04965842 In Healthy Male Subjects Using A 14c-microtracer Approach
Brief Title: Absorption, Metabolism, Excretion and Absolute Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7451008; 2017-000461-73 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-08-15 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Absorption, Metabolism, Excretion, Absolute Bioavailability
MeSH Terms: interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: This study will be an open label, non randomized, 2 period, fixed sequence, single dose study to characterize the absorption, metabolism and excretion of 14C- PF-04965842 and to evaluate the absolute oral bioavailability (F) and fraction absorbed (Fa) of PF-04965842 following oral administration of unlabeled PF-04965842 and IV and oral administration of 14C-PF-04965842 to healthy male subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mass Balance (Experimental): Cumulative recovery of radioactivity in urine and feces
  Interventions: Drug: PF-04965842
- Absolute Bioavailability (Experimental): Oral absolute bioavailability
  Interventions: Drug: Absolute Bioavailability

INTERVENTIONS:
Drug: PF-04965842 — 14C labeled PF-04965842
  Arms: Mass Balance
Drug: Absolute Bioavailability — Oral dose of unlabeled PF-04965842 and an IV dose of 14C labeled PF- 04965842
  Arms: Absolute Bioavailability

SUMMARY:
This study will investigate the absorption, metabolism and excretion of 14C-PF 04965842 and characterize plasma, fecal and urinary radioactivity and identify any metabolites, if possible, of 14C PF-04965842 in humans. In addition, this study will provide a better understanding of the pharmacokinetic disposition of PF-04965842 by obtaining intravenous (IV) clearance and delineating the extent of oral absorption (absolute bioavailability (F) and fraction absorbed (Fa)).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead electrocardiogram (ECG), or clinical laboratory tests.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with study confinement period, scheduled visits, treatment plan, laboratory tests, contraceptive requirements and other study procedures.

Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies).
2. Any clinically significant malabsorption condition (eg, gastrectomy, bowel resection).
3. A positive urine drug screen for drugs of abuse or recreational drugs.
4. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
5. History of abuse of alcohol or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 or more alcoholic drinks (male) in about 2 hours. As a general rule, alcohol intake should not exceed 21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
6. Use of tobacco/nicotine containing products in excess of 5 cigarettes/day.
7. Treatment with an investigational drug within 60 days.
8. Total 14C radioactivity measured in plasma exceeding 11 mBq/mL.
9. Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the blood pressure measurement should be repeated two more times and the average of the three measurements should be used to assess the subject's eligibility.
10. Supine 12 lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec at screening. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
11. Use of prescription or nonprescription drugs (including vitamins and dietary supplements) within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen may be used at doses of =<1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by Pfizer.
12. Use of herbal supplements within 28 days prior to the first dose of study medication.
13. Blood donation (excluding plasma donations) of no more than 100 mL or more within 56 days prior to dosing.
14. An estimated glomerular filtration rate of <90 mL/min/1.73 m2 based on the four variable Modification of Diet in Renal Disease (MDRD) equation.
15. History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON TB Gold test.
16. Any medical history of disease (ie, Gilbert's disease) that has the potential to cause a rise in total bilirubin over the upper limit of normal (ULN).
17. Subjects with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary:

    * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >=1.5 × ULN, total serum bilirubin >= 25.6 micromol/L;
    * Hemoglobin =<2.17 mmol/L (males).
18. Known participation in a clinical trial for PF 04965842 within 60 days prior to the first dose of study medication.
19. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
20. Unwilling or unable to comply with the Lifestyle Requirements described in this protocol.
21. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
22. Systemic therapy with any of the following medications that are CYP3A4 inhibitors within 7 days or 5 half lives (whichever is longer) or CYP3A inducers within 28 days prior to the first dose of the trial medication, or during the trial (Section 5.7).
23. History of sensitivity to heparin or heparin induced thrombocytopenia.
24. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
25. Subjects with conditions that affect their ability to taste ie, dysgeusia, respiratory infection, cold, etc.
26. Male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery of radioactivity | From predose to Day 14 day
  Total radioactivity in urine and feces based on total administered dose.

SECONDARY OUTCOMES:
Cmax | From predose to Day 5
  Maximum plasma concentration
Tmax | From predose to Day 5
  Time to maximum concentration
AUClast | From predose to Day 5
  Area under the plasma concentration-time curve from time 0 to last quantifiable concentration
AUCinf | From predose to Day 5
  Area under the plasma concentration-time curve from time zero to infinity
t1/2 | From predose to Day 5
  Apparent terminal elimination half-life
CL/F | From predose to Day 5
  Apparent total body clearance
Vz/F | From predose to Day 5
  Apparent volume of distribution
Vss (IV) | From predose to Day 5
  Steady State Volume of distribution
CL (IV) | From predose to Day 5
  Total Body Clearance
F | From predose to Day 5
  Absolute bioavailability= ratio of the adjusted geometric means of dose normalized AUCinf for unlabeled PF-04965842 and IV labeled 14C-PF-04965842
Fa | Predose to Day Day 5
  Fraction of PF 04965842 dose absorbed = Total 14C urine data following both IV and oral administration of 14C PF 04965842 (quantification by AMS).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bauman JN, Doran AC, King-Ahmad A, Sharma R, Walker GS, Lin J, Lin TH, Telliez JB, Tripathy S, Goosen TC, Banfield C, Malhotra BK, Dowty ME. The Pharmacokinetics, Metabolism, and Clearance Mechanisms of Abrocitinib, a Selective Janus Kinase Inhibitor, in Humans. Drug Metab Dispos. 2022 Aug;50(8):1106-1118. doi: 10.1124/dmd.122.000829. Epub 2022 Jun 14. PMID 35701182
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451008&StudyName=A+Phase+1%2C+Open-label%2C+Non-randomized%2C+2-period%2C+Fixed+Sequence%2C+Study+To+Investigate+The+Absorption%2C+Metabolism+And+Excretion+Of+%5B14c-pf-04965842%5D+And+To+Assess+The+Absolute+Bioavailability+And+Fraction+Absorbed+Of+Pf-04965842+In+Healthy+Male+Subjects+Using+A+14c+Microdose+Approach
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451008&StudyName=A+Phase+1%2C+Open-label%2C+Non-randomized%2C+2-period%2C+Fixed+Sequence+Study+To+Investigate+The+Absorption%2C+Metabolism+And+Excretion+Of+%5B14c-pf-04965842%5D+And+To+Assess+The+Absolute+Bioavailability+And+Fraction+Absorbed+Of+Pf-04965842+In+Healthy+Male+Subjects+Using+A+14c-microtracer+Approach